CLINICAL TRIAL: NCT02220777
Title: A Double-blind, Randomized, Placebo-controlled Study to Assess the Safety, Tolerability, Pharmacokinetics and Pharmacodynamics of Single Ascending Oral Doses of ASP8477 in Healthy Postmenopausal Females and Healthy Young Vasectomized Males, Including a Food Effect Part and a Part to Investigate the Interaction Between ASP8477 and Omeprazole
Brief Title: A Study to Assess the Effects of Single Ascending Doses (SAD) of ASP8477, the Effect That Food Has on the Drug, and the Interaction Between ASP8477 and Omeprazole in Healthy Postmenopausal Females and Healthy Young Vasectomized Males
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Europe B.V. (Industry)
Responsible Party: Sponsor
Organization: Astellas Pharma Inc (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: 8477-CL-0001; 2009-017865-42 (EudraCT Number)
Record Dates: First submitted 2014-08-18; First posted 2014-08-20 (Estimated); Last update posted 2014-08-20 (Estimated); Status verified 2014-08

CONDITIONS: Pharmacokinetics of ASP8477; Pharmacodynamics of ASP8477
Keywords: MTD (Maximum Tolerated Dose); Food effect; Postmenopausal subjects; Vasectomized subjects; FIH (First In Humans); SAD (Single Ascending Dose); DDI (Drug-Drug Interaction)
MeSH Terms: conditions — Metatropic dwarfism | interventions — ASP8477; Omeprazole

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1. ASP8477 and placebo (Experimental): Part 1: SAD in postmenopausal females and Part 2: SAD in vasectomized male
  Interventions: Drug: ASP8477; Drug: Placebo
- 2. ASP8477 alone (Experimental): Part 3, fasted or fed
  Interventions: Drug: ASP8477
- 3. omeprazole alone (Experimental): Part 4, Drug-Drug Interaction
  Interventions: Drug: omeprazole
- 4. ASP8477 + omeprazole (Experimental): Part 4: Drug-Drug Interaction
  Interventions: Drug: ASP8477; Drug: omeprazole

INTERVENTIONS:
Drug: ASP8477 — oral
  Arms: 1. ASP8477 and placebo; 2. ASP8477 alone; 4. ASP8477 + omeprazole
Drug: omeprazole — oral
  Arms: 3. omeprazole alone; 4. ASP8477 + omeprazole
Drug: Placebo — oral
  Arms: 1. ASP8477 and placebo

SUMMARY:
This is a 4-part study. Part I assesses the safety and tolerability of single ascending doses of ASP8477 or a placebo under fasted conditions in postmenopausal subjects. Part II is similar to part I except that the study is conducted in young, vasectomized males.

Part III assesses the effect of food (fed or fasted conditions) on ASP8477 in postmenopausal subjects.

Part IV assesses the drug-drug interaction between ASP8477 and omeprazole in postmenopausal subjects.

DETAILED DESCRIPTION:
Part I (SAD) in healthy postmenopausal females evaluates the safety, and tolerability, and defines Maximum Tolerated Dose = MTD, pharmacokinetics, and pharmacodynamics of single ascending oral doses (SAD) of ASP8477. It is anticipated that around 7 doses are required to cover the range from the safe starting dose until the MTD. Study medication is administered under fasted conditions. Based on the safety, PK, and clinical observation of the subjects, the dose escalation scheme may be adapted. Escalation to the next dose only proceeds after review of the safety, tolerability, and PK from the previous treatment period.

Part II (SAD in young, healthy, vasectomized males) is similar to Part I, one cohort of 12 subjects are treated with two doses of ASP8477 plus placebo. The doses tested depend on the safety data and pharmacodynamic profiles obtained in Part I, but is not expected to exceed MTD. The rationale for this part is to bridge the data obtained in female subjects to male subjects.

Part III (food effect) postmenopausal females receive ASP8477 once under fasted and once under fed conditions in two separate periods in random order. The dose does not exceed 1/3 of the MTD or, if that has not been reached, 1/3 of the highest tested dose in Part I. Subjects stay in the clinic for 2 periods of 5 to 7 days (depending on the terminal half life, resulting from Part I). Subjects are admitted on Day -2 per treatment period. Subjects' feeding status is the same as on Day 1 of the same treatment period. Subjects are given a single dose of ASP8477 under fed or fasting conditions on Day 1. After final discharge, subjects return for an End of Study Visit (ESV) 5-9 days later.

Part IV (ASP8477-omeprazole drug-drug interaction) postmenopausal subjects are randomized to receive omeprazole once alone and once with ASP8477 in two separate periods (in random order). The dose of ASP8477 is the MTD or, if that is not been reached, the highest tested dose in Part I. Omeprazole is chosen as target drug as it is a model substrate for CYP2C19 (accepted by FDA) and ASP8477 is known to have the strongest inhibitory effect on CYP2C19. Subjects are admitted on Day -1 and stay for 2 periods of 4 days. Subjects are given a single dose of omeprazole alone or with ASP8477 (in randomized order) on Day 1. Study medication is administered under fasted conditions. Subjects are discharged on Day 3 and return for an ESV 5-9 days later.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young (<65 years of age at first planned dose) postmenopausal female (Parts I, III, and IV).
* Healthy young vasectomized male subject aged 18-55 years inclusive (Part II).
* Body Mass index between 18.5 and 30.0 kg/m2 inclusive.

Exclusion Criteria:

* Known or suspected hypersensitivity to ASP8477 or any of the components of the formulations used.
* Any of the liver function tests above the upper limit of normal.
* A family history of psychiatric disorders.
* Use of grapefruit (more than 3 x 200 ml) or marmalade (more than three times) in the week prior to admission to the Clinical Unit, as reported by the subject.
* Use of xanthine-containing beverages within 48 hours before admission.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 72 (Actual)
Dates: Start 2010-11; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Safety as assessed by recording adverse events, physical examination, laboratory assessments, vital signs, electrocardiograms (ECGs), cortisol levels, arterial carbon dioxide and oxygen saturation | Day1 to End of Study Visit (5-9 days after final discharge)
  For Part I and II Bond-Lader Visual Analogue Scale (VAS) and Bowdle VAS assessments will also be taken.
The assessment of pharmacokinetic parameter of ASP8477 measured by Maximum concentration (Cmax), in plasma | Day 1 to Day 3
  Maximum concentration (Cmax)
The assessment of pharmacokinetic parameter of ASP8477 measured by Time to attain Cmax (tmax) in plasma | Day 1 to Day 3
  Time to attain Cmax (tmax)
The assessment of pharmacokinetic parameter of ASP8477 measured by Area Under the Curve (AUC) extrapolated until infinity (AUCinf) in plasma | Day 1 to Day 3
  Area Under the Curve (AUC) extrapolated until infinity (AUCinf)
The assessment of pharmacokinetic parameter of ASP8477 measured by AUC until last sample taken (AUClast) in plasma | Day 1 to Day 3
  AUC until last sample taken (AUClast), Absorption lag time (tlag), Apparent terminal elimination half-life (t1/2), Apparent volume of distribution (Vz/F), Apparent total body plasma clearance (CL/F)
The assessment of pharmacokinetic parameter of ASP8477 measured by Absorption lag time (tlag) in plasma | Day 1 to Day 3
  Absorption lag time (tlag)
The assessment of pharmacokinetic parameter of ASP8477 measured by Apparent terminal elimination half-life (t1/2) in plasma | Day 1 to Day 3
  Apparent terminal elimination half-life (t1/2)
The assessment of pharmacokinetic parameter of ASP8477 measured by Apparent volume of distribution (Vz/F) in plasma | Day 1 to Day 3
  Apparent volume of distribution (Vz/F)
The assessment of pharmacokinetic parameter of ASP8477 measured by Apparent total body plasma clearance (CL/F) in plasma | Day 1 to Day 3
  Apparent total body plasma clearance (CL/F)
The assessment of pharmacokinetic parameter of ASP8477 measured by Amount excreted in urine until last sample (Aelast) in urine | Day 1 to Day 3
  Amount excreted in urine until last sample (Aelast)
The assessment of pharmacokinetic parameter of ASP8477 measured by Cumulative amount of unchanged drug excreted into the urine from time zero to infinity after single dose (Aeinf) in urine | Day 1 to Day 3
  Cumulative amount of unchanged drug excreted into the urine from time zero to infinity after single dose (Aeinf)
The assessment of pharmacokinetic parameter of ASP8477 measured by Percentage of unchanged drug excreted into the urine from time of last measurable concentration (Aelast%) in urine | Day 1 to Day 3
  Percentage of unchanged drug excreted into the urine from time of last measurable concentration (Aelast%)
The assessment of pharmacokinetic parameter of ASP8477 measured by Percentage of unchanged drug excreted into the urine from time zero to infinity after single dose (Aeinf%) in urine | Day 1 to Day 3
  Percentage of unchanged drug excreted into the urine from time zero to infinity after single dose (Aeinf%)
The assessment of pharmacokinetic parameter of ASP8477 measured by Renal clearance (CLR) in urine | Day 1 to Day 3
  Renal clearance (CLR)

SECONDARY OUTCOMES:
The assessment of pharmacokinetics of omeprazole measured by plasma concentration | Day 1 to Day 3
  Cmax, tmax, AUCinf, AUClast, t1/2, Vz/F, CL/F
The assessment of pharmacodynamics of ASP8477 measured by serum concentration | Day 1 to Day 4
  serum concentration of endogenous substrates, volume of urine production, GFR and intra-ocular pressure

CONTACTS AND LOCATIONS:
Overall Officials: Study Manager, Study Chair — Astellas Pharma Europe B.V.
Locations (2):
- SGS Belgium N.V., Antwerp, Belgium
- SGS Aster, Paris, France